CLINICAL TRIAL: NCT01778868
Title: Endocrine Disrupting Environmental Chemicals: From Accumulation to Their Role in the Global "Neuro-endocrine" Epidemic of Obesity and Its Metabolic Consequences
Brief Title: Environmental Chemicals and Their Role in Obesity
Acronym: ENDORUP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Ethisch Comité UZ Antwerpen, Ethisch Comité UZ Antwerpen, University Hospital, Antwerp
Other Study IDs: ENDORUP
Record Dates: First submitted 2013-01-18; First posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples Urinary samples Fat samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Overweight and obese individuals
- Normal weight individuals

SUMMARY:
Hormonal disruption is the inappropriate alteration of the hormonal system by chemical substances that are present in our environment. Some chemical substances are capable of replicating, enhancing or reducing the production, release, transport or action of natural hormones. Therefore, they are called hormonal or endocrine disrupters. Some 'classic' endocrine disrupters such as pesticides and dioxins are considered responsible for infertility, cancer and thyroid problems. Recently, a number of additional chemical substances were stipulated to have endocrine disrupting capabilities. The industrial production of these substances in large quantities has led to an accumulation in our environment and thus possible negative consequences on human health.

The aim of this study is to investigate the rol of these chemical substances in the occurence of overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* adult
* Overweight (BMI > 25 kg/m²) or obesity (BMI > 30 kg/²)

Exclusion Criteria:

* Type 1 diabetes mellitus
* psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with BMI > 25kg/m² and a normal weight (BMI < 25 kg/m²) control population
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2009-08; Primary Completion 2013-03 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Serum levels of polychlorinated biphenyls | at the moment of entering a weight loss program
  The following PCB congeners are measured (official IUPAC number is given):
  CB 28 CB 52 CB 74 CB 95 CB 99 CB 101 CB 105 CB 118 CB 149 CB 146 CB 153 CB 138 CB 187 CB 183 CB 128 CB 167 CB 174 CB 177 CB 171 CB 172 CB 156 CB 180 CB 170 CB 199 CB 196/203 CB 194 CB 206 CB 209
Serum levels of hydroxylated metabolites of polychlorinated biphenyls | at the moment of entering a weight loss program
  The following hydroxylated metabolites of polychlorinated biphenyls are measured 4-HO-CB79 4-HO-CB120 3HO-CB118 4HO-CB107 3HO-CB153 4HO-CB146 4HO-CB127 3HO-CB138 4HO-CB130 4HO-CB163 4HO-CB187 4-HO-CB162 4-HO-CB177 3HO-CB180 4HO-CB172 4HO-CB193 4-diMeO-CB202 4-HO-CB208
serum levels of organochlorine pesticides | at the moment of entering a weight loss program
  The following organochlorine pesticides are measured:
  alfa- hexachlorocyclohexane, beta-hexachlorocyclohexane, gamma-hexachlorocyclohexane Hexachlorobenzen Ocychlordane Transnonachlor p-p-dichlorodiphenyltrichloroethane, p,p'-dichlorodiphenyldichloroethylene pp-dichlorodiphenyldichloroethane
serum levels of polybrominated diphenyl ethers | at the moment of entering a weight loss program
  The following polybrominated diphenyl ethers (BDE) are measured: BDE 28 BDE 47 BDE 100 BDE 99 BDE 154 BDE 153 BDE 183
Urinary levels of pollutants | at the moment of entering a weight loss program
  The pollutants detected in urine comprise of bisphenol A, triclosan, phtalates
Change in serum levels of polychlorinated biphenyls compared to the levels at the start of the weight loss program | after 3, 6 and 12 months of weight loss
  The following PCB congeners are measured (official IUPAC number is given):
  CB 28 CB 52 CB 74 CB 95 CB 99 CB 101 CB 105 CB 118 CB 149 CB 146 CB 153 CB 138 CB 187 CB 183 CB 128 CB 167 CB 174 CB 177 CB 171 CB 172 CB 156 CB 180 CB 170 CB 199 CB 196/203 CB 194 CB 206 CB 209
change in serum levels of hydroxylated metabolites of polychlorinated biphenyls compared to the level at the start of the weight loss program | after 3,6 and 12 months of weigth loss
  The following hydroxylated metabolites of polychlorinated biphenyls are measured 4-HO-CB79 4-HO-CB120 3HO-CB118 4HO-CB107 3HO-CB153 4HO-CB146 4HO-CB127 3HO-CB138 4HO-CB130 4HO-CB163 4HO-CB187 4-HO-CB162 4-HO-CB177 3HO-CB180 4HO-CB172 4HO-CB193 4-diMeO-CB202 4-HO-CB208
Change in serum levels of organochlorine pesticides compared to the level at the start of the weight loss program | after 3,6 and 12 months of weight loss
  The following organochlorine pesticides are measured:
  alfa- hexachlorocyclohexane, beta-hexachlorocyclohexane, gamma-hexachlorocyclohexane Hexachlorobenzen Ocychlordane Transnonachlor p-p-dichlorodiphenyltrichloroethane, p,p'-dichlorodiphenyldichloroethylene pp-dichlorodiphenyldichloroethane
Change in serum levels of polybrominated diphenyl ethers compared to the level at the start of the weight loss program | After 3,6 and 12 months of weight loss
  The following polybrominated diphenyl ethers (BDE) are measured: BDE 28 BDE 47 BDE 100 BDE 99 BDE 154 BDE 153 BDE 183
change in urine levels of pollutants compared to the level at the start of the weight loss program | after 3,6 and 12 months of weight loss
  The pollutants detected in urine comprise of bisphenol A, triclosan, phtalates

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Jorens, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerpen, Belgium

REFERENCES:
- [Derived] Dirinck EL, Dirtu AC, Govindan M, Covaci A, Jorens PG, Van Gaal LF. Endocrine-disrupting polychlorinated biphenyls in metabolically healthy and unhealthy obese subjects before and after weight loss: difference at the start but not at the finish. Am J Clin Nutr. 2016 Apr;103(4):989-98. doi: 10.3945/ajcn.115.119081. PMID 26961932
- [Derived] Dirinck E, Dirtu AC, Jorens PG, Malarvannan G, Covaci A, Van Gaal LF. Pivotal Role for the Visceral Fat Compartment in the Release of Persistent Organic Pollutants During Weight Loss. J Clin Endocrinol Metab. 2015 Dec;100(12):4463-71. doi: 10.1210/jc.2015-2571. Epub 2015 Oct 15. PMID 26469381
- [Derived] Dirinck EL, Dirtu AC, Govindan M, Covaci A, Van Gaal LF, Jorens PG. Exposure to persistent organic pollutants: relationship with abnormal glucose metabolism and visceral adiposity. Diabetes Care. 2014 Jul;37(7):1951-8. doi: 10.2337/dc13-2329. PMID 24963112